CLINICAL TRIAL: NCT03065400
Title: PD-1 Inhibition in Advanced Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Massachusetts General Hospital (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2350
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Chronic Phase Myelofibrosis; Primary Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Polycythemia Vera
Keywords: Myelofibrosis; Acute Leukemia
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg of Pembolizumab administered via intravenous infusion over 30 mins given every 3 weeks
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to test the effectiveness of a drug called pembrolizumab in patients with Myeloproliferative Neoplasm (MPN); chronic phase (MF-CP), accelerated phase (MPN-AP), or blast phase (MF-BP). Myelofibrosis neoplasm (MPN) is a group of diseases of the bone marrow in which excessive cells are produced.

Pembrolizumab also known as Keytruda is a drug that has recently been approved in the United Stated by the Food and Drug Administration (FDA) for the treatment of patients with unresectable or metastatic melanoma and disease progression. Pembrolizumab is experimental in the treatment of MPN. The researchers want to find out what effects, good and /or bad it has on participants and the disease.

Participants qualify to take part in this research study if have been diagnosed with a MPN blood disorder called myelofibrosis (MF). Accelerated (10-19% blasts in the blood or bone marrow) and blast phase (>20% blasts in the blood or bone marrow) MPN has been a difficult disease to treat. The term "blasts" refers to immature cells found in the bone marrow. They are not fully developed, and therefore, do not yet carry out any particular function within the body.

Funds for conducting this research are provided by Merck and Company, the manufacturer of the study drug pembrolizumab.

DETAILED DESCRIPTION:
The researchers propose a Simon-two stage design for this study. The researchers will test pembrolizumab at the FDA approved dose (in head and neck cancer) of 200mg dose administered via intravenous infusion over 30 minutes given every 3 weeks. Nine patients will be enrolled in the first stage of the Simon-two stage design, and 15 in the second stage. A treatment cycle is 3 weeks and the core study period is 6 cycles. Response assessment by established consensus criteria will be used to assess response after 6 cycles in order to determine if the trial will progress to the second stage and for the purpose of determining the primary endpoint. In addition, allowed will be a maximum of ten patients with accelerated or blast phase disease (MPN-AP/BP) who are refractory or intolerant to conventional therapies such as decitabine, and in which hematopoietic stem cell transplant is not a therapeutic option (exploratory cohort), to enroll in the study as a separate exploratory cohort. These patients can be enrolled during stage 1 or 2 and will be analyzed separately from the primary cohort population.

Exploratory biomarkers will be obtained from enrolled patients at baseline, cycle 3 and cycle 7 and at 1 year of therapy. Patients that obtain at least a clinical improvement after 6 cycles of therapy can continue receiving pembrolizumab until evidence of disease progression, unacceptable toxicity, and patient or physician decision for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing consent.
* Must have a diagnosis of chronic phase (CP) (defined as peripheral blood and bone marrow <10% blasts) primary myelofibrosis (PMF) or post essential thrombocythemia (post-ET) or polycythemia vera (post-PV) myelofibrosis by World Health Organization (WHO) criteria OR a diagnosis of a myeloproliferative neoplasm in accelerated/blast phase (MPN-AP/BP) defined as either a peripheral blood or bone marrow with =10% blasts .
* If the diagnosis is MF-CP, must have Dynamic International Prognostic Scoring System (DIPSS) intermediate-2/high risk disease and either be intolerant/resistant to ruxolitinib as determined by the treating investigator or ineligible for ruxolitinib therapy as determined by the treating investigator .
* If the diagnosis is MPN-AP/BP, must have progressive/resistant disease after treatment with a DNMT1 inhibitor therapy (azacytidine, decitabine) as determined by the treating investigator .
* Either not eligible or unwilling to proceed with hematopoietic stem cell transplantation (HSCT)
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., = Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., = Grade 1 or at baseline) from adverse events due to a previously administered agent.

  1. Note: Subjects with = Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. "Anti-CD137 or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Gabriela Hobbs, MD, Study Chair — Harvard Medical School Massachussets General Hospital
Locations (3):
- United States (3):
  - Harvard Medical School Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center Division of Hematology, Department of Oncology, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hobbs G, Cimen Bozkus C, Moshier E, Dougherty M, Bar-Natan M, Sandy L, Johnson K, Foster JE, Som T, Macrae M, Marble H, Salama M, El Jamal SM, Zubizarreta N, Wadleigh M, Stone R, Bhardwaj N, Iancu-Rubin C, Mascarenhas J. PD-1 inhibition in advanced myeloproliferative neoplasms. Blood Adv. 2021 Dec 14;5(23):5086-5097. doi: 10.1182/bloodadvances.2021005491. PMID 34581778

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembolizumab: 200 mg of Pembolizumab administered via intravenous infusion over 30 mins given every 3 weeks
Period: Overall Study
Arm/Group | Pembolizumab
Started | 10
Completed | 0
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1
Not completed — Completed 6 cycles but did not meet criteria to continue past cycle 6 | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pembolizumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 70 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: European Leukemia Net -International Working Group (ELN-IWG) Criteria
Description: The proportion of treated MF-CP patients (primary cohort) that achieve at least a clinical improvement (CI, PR, CR) by combined European Leukemia Net -International Working Group (ELN-IWG) criteria after 6 cycles of pembrolizumab therapy.
  Complete Remission - CR: Bone marrow: Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF and Peripheral blood: Hemoglobin ≥100 g/L and <UNL; neutrophil count ≥ 1 × 109/L and <UNL; Platelet count ≥100 × 109/L and <UNL; <2% immature myeloid cells and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH Partial Remission (PR): Hemoglobin ≥100 g/L and <UNL; neutrophil count ≥1 × 109/L and <UNL; platelet count ≥100 × 109/L and <UNL; <2% immature myeloid cells and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH or Bone marrow: Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF, and Hemoglobin ≥85 but <100 g/L and <UNL; neutrophil count ≥1 × 109/L and <UNL; plat
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembolizumab
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Acute Myeloid Leukemia Response Criteria
Description: The proportion of treated MPN-AP/BP patients (exploratory cohort) that achieve at least a complete morphologic remission of the leukemic blasts (CR, Cri) by Acute Myeloid Leukemia Response Criteria within 6 cycles of pembrolizumab therapy.
  Acute Myeloid Leukemia Response Assessment Criteria:
  Complete Response (CR) - The subject must be free of all symptoms related to leukemia and have an absolute neutrophil count of greater than 1 x 109/L, no need for red blood cell transfusion, platelet count greater than 100x 109/L, and normal marrow differential (<5% blasts) in a normo- or hypercellular marrow Complete Remission with Incomplete Hematologic Recovery (Cri) - As per CR but incomplete count recovery Partial Response - CR with 6-25% abnormal cells in the marrow or 50% decrease in bone marrow blasts
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembolizumab
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Pembolizumab
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembolizumab (N=10)
Weakness (Nervous system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
High grade pleomorphic sarcoma of left breast. (Reproductive system and breast disorders) | 1
Respiraitory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembolizumab (N=10)
Anemia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 5
WBC Decreeased (Blood and lymphatic system disorders) | 4
AST Increased (Hepatobiliary disorders) | 3
Hyperglycemia (Endocrine disorders) | 5
Hyperuricemia (Renal and urinary disorders) | 4
Hypoalbuminemia (Hepatobiliary disorders) | 3
ALP Increased (Hepatobiliary disorders) | 2
Hypocalcaemia (Renal and urinary disorders) | 2
Hypernatremia (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Fatigue (General disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Fever (General disorders) | 3
Headache (Nervous system disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Weakness (Nervous system disorders) | 3
Blurred Vision (Nervous system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2
Weight Loss (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03065400/Prot_SAP_000.pdf